CLINICAL TRIAL: NCT06146478
Title: Deciphering Effects of Thalidomide on Red Blood Cells in Transfusion Dependents Beta Thalassemia Patients: A Pharmacodynamics and Pharmacogenetics Analysis
Brief Title: Deciphering Effects of Thalidomide on Red Blood Cells in Transfusion Dependents Beta Thalassemia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blood Care Clinic (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Inayat ur Rahman, PhD Scholar, Blood Care Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dir/KMU-EB/TC/000863
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Transfusion-dependent Beta-Thalassemia
Keywords: β-thalassemia; Thalidomide; β- globin mutations; Single Nucleotide Polymorphisms
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Intervention Model Description: Patients will be grouped into thalidomide and non-thalidomide groups on the basis of their willingness to receive thalidomide therapy. Thalidomide will be given at an average dose of 1.5mg/kg/day (range 1-2mg/kg/day). Patients will be followed up for 12 months and data will be collected at different visits.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thalidomide Group (Experimental): In addition to routine β-thalassemia treatment patients in this group also received thalidomide at an average dose of 1.5mg/kg/day
  Interventions: Drug: Thalidomide
- Non-Thalidomide Group (No Intervention): Participants received routine treatment for β-thalassemia such as regular blood transfusion and hydroxyurea at an average dose of 20mg/kg/day

INTERVENTIONS:
Drug: Thalidomide — Thalidomide given at an average dose of 1.5mg/kg/day
  Other Names: Bludomide
  Arms: Thalidomide Group

SUMMARY:
The goal of this Non-Randomized Clinical Trial is to determine the effects of thalidomide on red blood cells in transfusion dependent beta thalassemia patients. The main aims of this study are:

* To determine the therapeutic effect of Thalidomide on hemoglobin.
* To analyze association of different β- globin mutations with response to thalidomide in β-thalassemia patients.
* To analyze association of Single Nucleotide Polymorphisms (SNPS) of HBG2, BCL11A and HBS1L-MYB with response to thalidomide in β-thalassemia patients.
* To correlate GATA1 and KLF1 gene expression with response to thalidomide in β-thalassemia patients.

Patients will be grouped into thalidomide and non-thalidomide groups on the basis of their willingness to receive thalidomide therapy. Thalidomide will be given at an average dose of 1.5mg/kg/day (range 1-2mg/kg/day). Patients will be followed up for 12 months and data will be collected at different visits. After 12 months of thalidomide therapy patients will be divided into responders and non-responders for comparative analyses on the basis of increase in hemoglobin level.

DETAILED DESCRIPTION:
Thalassemias are a group of genetic disorder of hemoglobin synthesis characterized by a decreased synthesis of globin chain. Thalassemias are classified as α-,β-, γ-,or δ-thalassemias depending upon the chain whose synthesis is reduced. Among these, β-thalassemia is more common. In β-thalassemia there is a decreased or absent hemoglobin A (HbA). Normal adult hemoglobin is primarily HbA, which represents approximately 98% of circulating hemoglobin. HbA is formed from 2 α and 2 β chains (α2β2). Combination of 2 α and 2 δ (α2δ2) form hemoglobin A2 (HbA2). Combination of 2 α and 2 γ (α2γ2) form hemoglobin F (HbF) which is a major form of hemoglobin in fetal life but comprises less than 1% of adult hemoglobin. Human beta-globin protein is encoded by HBB gene on chromosome 11, which contributes two β polypeptide chains. Therefore, one chain is inherited from the mother and one inherited from the father. In normal (homozygote) both genes are normal and produce normal β polypeptide chains to normal quantity. In heterozygote one gene is normal and other is abnormal which does not produce β polypeptide chain. Such condition is called β-thalassemia minor. In such a person normal gene produces enough β chain to maintain hemoglobin level. In abnormal homozygote both beta chain genes are abnormal and do not produce β polypeptide chain. Such condition is called β-thalassemia major. Reduced or absent production of β-globin chains with relative excess of α-chains cause imbalance and free α chains precipitate within the red blood cells. This result in extensive premature destruction of red cell precursors in the bone marrow, referred to as "ineffective erythropoiesis". The imbalance causes peripheral hemolysis as well. The two phenomena culminate in clinically significant anemia.

Severity of anemia due to β-thalassemia depends upon the type of mutations in β-globin gene. Mostly point mutations and frame shift mutations, in intronic as well exonic region, are reported in Pakistani β-thalassemia patients. Some mutations completely block the β-gene and thus no β globin chain is produced (βo) while in other mutations there is production of some β globin chains (β+). In β-thalassemia major both β globin alleles undergo mutations (βo/βo) and disease is severe. In β-thalassemia minor only one of β globin alleles are mutated (β+/β or βo/β) and patient is asymptomatic. β-thalassemia intermedia (β+/β+ or βo/β+) is the form of disease which is milder than thalassemia major but more severe than thalassemia minor. Besides less severe β+ mutations, inheritance of HbF inducing genetic variations and co-inheritance of alpha globin mutations can also ameliorate the clinical severity of the disease. In regards to HbF induction, genetic association studies have shown that there are at least three major loci that play a major role in increasing HbF and are associated with severity of β-thalassemia. These include -158 C > T in the promoter gene Gamma 2 (locus XmnI), intergenic regions HBS1L-MYB in the 6q23.3 chromosomal region, and the BCL11A gene on chromosome 2p16.1.

Annually about 60000 babies are born with thalassemia all over the world. Global annual incidence of β-thalassemia is estimated at a rate of 1/100,000 . Carrier rate for β-thalassemia in Pakistan ranges between 5-8%, and around 5000 children are diagnosed each year with the disease .

Severe anemia in β-thalassemia patients necessitates frequent transfusions, which lead to iron overload. Chronic anemia and iron overload lead to several complications including skeletal deformities, splenomegaly, osteoporosis, endocrinopathies, growth retardation and cardiac complications. Iron overload is treated with iron chelating agents. Definitive treatment is bone marrow transplantation (9).Thalassemia patients who do not respond well to blood transfusions can take hydroxyurea or thalidomide, and sometimes a combination of both.

Thalidomide, an immuno-modulatory drug is currently approved by FDA for the treatment of multiple myeloma and Leprosy. Thalidomide is used off-label for the treatment of β-thalassemia patients worldwide. Thalidomide has been reported to reduce or even eliminate the need for red blood cell transfusions in patients with transfusion dependent β-thalassemia . Although association of β globin gene mutations and genetic modifiers with severity of β-thalassemia have been well studied but association of these genetic factors with response to thalidomide therapy still needs to be explored. A study conducted on 48 Chinese patients showed association of Xmn1 HBG2, BCL11A & HBSIL-MYB single nucleotide polymorphisms (SNPs) with response to thalidomide therapy. .

Improved terminal erythroid maturation and red blood cells stability are considered effective therapeutic approaches in the treatment of thalassemia. GATA1 and KLF1 are important transcription factor in erythroid differentiation which play critical role in regulation of globin gene expression. Studies reveal that increased expression of GATA1 and KLF1 causes induction of fetal hemoglobin (HbF) leading to reduced accumulation of α-globin chains in erythroid precursors and betterment of imbalance between α and β chains thus diminished ineffective erythropoiesis.

The current study aims to determine the in-vivo effects of thalidomide on GATA1 & KLF1 gene expression in transfusion dependent β-thalassemia patients. Findings of the study will provide scientific evidence in support or against the off- label use of thalidomide in β-thalassemia patients. Results of the study regarding association of β-globin mutations and Xmn1 HBG2 BCL11A & HBSIL-MYB single nucleotide polymorphisms with response to thalidomide therapy will explain variation in inter-individual response to the drug and thus help in predicting response before starting thalidomide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed transfusion dependent β-thalassemia patients
* Possess a verified pre transfusion Hb electrophoresis report performed at age≥ 6 months

Exclusion Criteria:

* Patients with active metabolic or systemic comorbidities
* Patients with autologous antibodies, AIHA or hypersplenism

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Response to thalidomide on the basis of increase in hemoglobin (Hb) level at 12 months of treatment. | Baseline, 1 month, 6 months and 12 months
  On the basis of increase in Hb level patients categorized as follows:
  1. Excellent Responders (ER): In whom the Hb level raised to ≥9.0g/dl without any transfusion in the last two months.
  2. Good Responders (GR): In whom the Hb level raised to 7.0-8.9 g/dL without any transfusion in the last two months.
  3. Partial Responders (PR): In whom the Hb level remained <7.0 g/dL but did raise to a significantly higher level than the base-line without any transfusion in the last two months.
  4. Non-Responders (NR): In whom the Hb level did not show any significant improvement in comparison to the base-line
Association of different β- globin mutations with response to thalidomide | Baseline
  Amplification refractory mutation system polymerase chain reaction (ARMS-PCR) is used for detection of β- globin mutations.
Association of Single Nucleotide Polymorphisms (SNPS) of HBG2, BCL11A and HBS1L-MYB with response to thalidomide | Baseline
  PCR & DNA Sequencing are used for SNP genotyping

SECONDARY OUTCOMES:
Change from baseline in GATA1 and KLF1 gene expression at 12 months of thalidomide treatment | Baseline and after 12 months
  Real Time-Polymerase Chain Reaction (RT-PCR) is used for analysis of gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Sami Siraj, PhD, Study Director — Institute Of Pharmaceutical Sciences, Khyber Medical University Peshawar
Locations (1):
- Blood Care Clinic, Peshawar, Khyber Pakhtunkhwa, Pakistan

REFERENCES:
- [Background] Ren Q, Zhou YL, Wang L, Chen YS, Ma YN, Li PP, Yin XL. Clinical trial on the effects of thalidomide on hemoglobin synthesis in patients with moderate thalassemia intermedia. Ann Hematol. 2018 Oct;97(10):1933-1939. doi: 10.1007/s00277-018-3395-5. Epub 2018 Jun 22. PMID 29931453
- [Background] Aerbajinai W, Zhu J, Gao Z, Chin K, Rodgers GP. Thalidomide induces gamma-globin gene expression through increased reactive oxygen species-mediated p38 MAPK signaling and histone H4 acetylation in adult erythropoiesis. Blood. 2007 Oct 15;110(8):2864-71. doi: 10.1182/blood-2007-01-065201. Epub 2007 Jul 9. PMID 17620452
- [Background] Yang K, Wu Y, Ma Y, Xiao J, Zhou Y, Yin X. The association of HBG2, BCL11A, and HBS1L-MYB polymorphisms to thalidomide response in Chinese beta-thalassemia patients. Blood Cells Mol Dis. 2020 Sep;84:102442. doi: 10.1016/j.bcmd.2020.102442. Epub 2020 Apr 26. PMID 32387854
- [Background] Ehnert S, Linnemann C, Braun B, Botsch J, Leibiger K, Hemmann P, Nussler AAK. One-Step ARMS-PCR for the Detection of SNPs-Using the Example of the PADI4 Gene. Methods Protoc. 2019 Jul 25;2(3):63. doi: 10.3390/mps2030063. PMID 31349745
- [Background] Grzasko N, Chocholska S, Goracy A, Hus M, Dmoszynska A. Thalidomide can promote erythropoiesis by induction of STAT5 and repression of external pathway of apoptosis resulting in increased expression of GATA-1 transcription factor. Pharmacol Rep. 2015 Dec;67(6):1193-200. doi: 10.1016/j.pharep.2015.05.011. Epub 2015 May 29. PMID 26481541
- [Background] Martinez PA, Li R, Ramanathan HN, Bhasin M, Pearsall RS, Kumar R, Suragani RNVS. Smad2/3-pathway ligand trap luspatercept enhances erythroid differentiation in murine beta-thalassaemia by increasing GATA-1 availability. J Cell Mol Med. 2020 Jun;24(11):6162-6177. doi: 10.1111/jcmm.15243. Epub 2020 Apr 29. PMID 32351032
- [Background] Jalali Far MA, Dehghani Fard A, Hajizamani S, Mossahebi-Mohammadi M, Yaghooti H, Saki N. Thalidomide is more efficient than sodium butyrate in enhancing GATA-1 and EKLF gene expression in erythroid progenitors derived from HSCs with beta-globin gene mutation. Int J Hematol Oncol Stem Cell Res. 2016 Jan 1;10(1):37-41. PMID 27047649
- [Background] Guillem F, Dussiot M, Colin E, Suriyun T, Arlet JB, Goudin N, Marcion G, Seigneuric R, Causse S, Gonin P, Gastou M, Deloger M, Rossignol J, Lamarque M, Choucair ZB, Gautier EF, Ducamp S, Vandekerckhove J, Moura IC, Maciel TT, Garrido C, An X, Mayeux P, Mohandas N, Courtois G, Hermine O. XPO1 regulates erythroid differentiation and is a new target for the treatment of beta-thalassemia. Haematologica. 2020 Sep 1;105(9):2240-2249. doi: 10.3324/haematol.2018.210054. PMID 33054049
- [Background] Yang K, Wu Y, Zhou Y, Long B, Lu Q, Zhou T, Wang L, Geng Z, Yin X. Thalidomide for Patients with beta-Thalassemia: A Multicenter Experience. Mediterr J Hematol Infect Dis. 2020 May 1;12(1):e2020021. doi: 10.4084/MJHID.2020.021. eCollection 2020. PMID 32395210
- [Derived] Rahman IU, Khan MTM, Ali Z, Ahmad S, Shahid M, Zafar S, Aamir FF, Khan I, Ali M, Jelani M, Khan K, Ahmad N, Yousafzai Y, Mian AA, Siraj S. Thalidomide confers therapeutic benefit in beta thalassemia patients by enhancing hemoglobin and hematopoietic gene expression: A non-randomized clinical trial. Blood Cells Mol Dis. 2025 Jul-Sep;113-114:102936. doi: 10.1016/j.bcmd.2025.102936. Epub 2025 May 23. PMID 40446669